CLINICAL TRIAL: NCT03287375
Title: Treatment of Peritoneal Carcinomatosis With Pressurized IntraPeritoneal Aerosol - The PIPAC-OPC2 Trial
Brief Title: Treatment of Peritoneal Carcinomatosis With Pressurized IntraPeritoneal Aerosol Chemotherapy -
Acronym: PIPAC-OPC2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-OPC2
Record Dates: First submitted 2017-09-02; First posted 2017-09-19 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Peritoneum; Carcinomatosis; Peritoneal Neoplasms; Peritoneal Metastases; Chemotherapy Effect; Chemotherapeutic Toxicity; Quality of Life; Histologic Progression
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — Cisplatin; Doxorubicin; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Cohorte study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIPAC (Experimental): Peritoneal metastases (PM) from colorectal or appendiceal cancer will be treated with Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) using oxaliplatin 92 mg/m2 in 150 ml dextrose. Peritoneal metastases (PM) from other GI or gynecologic cancers will be treated with Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) using cisplatin 7.5 mg/m2 in 150 ml saline combined with doxorubicin 1.5 mg/m2 in 50 ml saline. PIPAC is performed during a standard laparoscopy with a capnoperitoneum of 12 mmHg and the aerosolised chemotherapy will be nebulized at a maximum pressure of 200 PSI and a flow rate of 0.5 ml/min. There is no upper number of allowed PIPAC treatments, but they will be planned in series of 3 with 4-6 weeks interval (6-7 weeks if combined with systemic chemotherapy).
  Interventions: Drug: PIPAC

INTERVENTIONS:
Drug: PIPAC
  Other Names: Cisplatin; Doxorubicin; Oxaliplatin

SUMMARY:
This is a study, where the efficacy of Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) against peritoneal metastases will be evaluated. Furthermore, this study will focus on the best evaluation method, where both Quality of Life questionnaires, repeated histology, cytology and MRI will be used.

DETAILED DESCRIPTION:
Patients with peritoneal metastases (PM) will be reviewed by the interdisciplinary tumor board and included based on predefined in- and exclusion criteria. Eligible candidates with primary colorectal or appendiceal cancers will be treated with intraperitoneal oxaliplatin delivered by the PIPAC procedure, while patients with other primary cancers will be treated with a combination of cisplatin and doxorubicin. Three PIPAC treatments will be scheduled in intervals of 4-6 weeks (6-7 if combined with systemic chemotherapy). MRI and QoL questionnaires will be performed at baseline and after three PIPAC treatments. If the patients respond to the PIPAC treatment, further courses of PIPAC can be planned at the tumour board meeting.

In brief, PIPAC is performed during a standard laparoscopy using two access ports, where the magnitude of PM is evaluated using the Peritoneal Carcinosis Index and the Dutch 7 regions count. Afterwards, the peritoneum is biopsied at different regions and peritoneal lavage fluid is sent for cytology. Then, chemotherapy is aerosolised within the abdomen, and after 30 minutes, the aerosol has been absorbed by the peritoneum, and the patient is closed according to departmental guidelines. The patients are expectedly discharged within 24 hours, and will after each PIPAC treatment be screened for adverse events using the CTCAE and Dindo-Clavien classification.

Amendment 23-03-2020:

Title Evaluation of the Peritoneal Regression Grading Score in biopsies from clips marked peritoneal metastases compared to biopsies from the element with most malignant features during repeated Pressurized IntraPeritoneal Aerosol Chemotherapy

Background Patients with peritoneal metastases (PM) may be treated with protocolled Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) at Odense PIPAC Center by inclusion in the prospective PIPAC-OPC2 study. The response evaluation is based on repeated biopsies from clips marked PM elements retrieved during each PIPAC procedure. Histological regression is categorized by the Peritoneal Regression Grading Score (PRGS). While the PRGS is internationally validated and accepted, there is a lack of consensus regarding the biopsy strategy during subsequent PIPAC procedures. As part of the PIPAC-OPC2 protocol, we define the element with most malignant features in each of the four abdominal quadrants during the first PIPAC procedure. We clips mark these elements to be able to take biopsies from the same area during subsequent procedures, thus reducing sampling error. At other centres, the biopsies are taken from those elements that are most suspicious of malignancy at visual inspection during each PIPAC.

The question is whether the histological regression in repeated biopsies from clips marked elements is influenced by fibrosis from the clips or dominated by scar tissue induced by the biopsy per se. Moreover, it is possible that PMs may progress in unmarked areas, in spite of regression in the marked areas. Hypothetically, this could lead to false positive regression, thus overestimating the histological response to PIPAC.

Objective To investigate if the histologically assessed response to PIPAC is dependent on the biopsy strategy: Biopsies taken from those areas that are most suspicious of malignancy at visual inspection compared to re-biopsies of the same, clips marked PM elements during the second PIPAC procedure.

Number of patients Data from 131 consecutive patients included in the PIPAC-OPC1 or PIPAC-OPC2 studies show that 67% had more than one PIPAC procedure. The mean PRGS was reduced by 0.38 points (SD 0.65) from PIPAC 1 to PIPAC 2, based on re-biopsies from clips marked elements.

With an alpha of 0.05 and a power of 0.80, 25 patients are needed to test the null hypothesis of no difference between the two biopsy strategies. Patients are their own control.

Methods The present study is an amendment to the PIPAC-OPC2 study. To date, 101/137 patient have been included. With an expected study termination of no more than 30% of the patients before PIPAC 2, this amendment is feasible within the framework of the PIPAC-OPC2 study.

A clips marked element is defined as the area covered within two times the length of the opened jaws of a biopsy forceps. An external surgical oncologist with vast experience of staging cancer patients will define the PM element with most malignant features before retrieval of biopsies during the second PIPAC procedure. Accordingly, biopsies will then be taken from the clips marked elements and the defined element with most malignant features (potentially same element). The pathologist will be blinded during the analyses of biopsies from the second PIPAC procedure.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological verified gastrointestinal-, ovarian- or primary peritoneal malignancy (based on tissue from the primary tumor and/or its metastases).
* Ovarian cancer patients must be platinum resistant and have completed at least one line of chemotherapy for platinum resistant disease.
* Radiological, histological or cytological evidence of PC.
* No indication for CRS and HIPEC (according to National Guidelines).
* Performance status 0-1.
* No more than a single extra-peritoneal metastasis.
* Age > 18 years.
* Females must be post-menopausal
* Written informed consent must be obtained according to the local Ethics Committee requirements.

Exclusion Criteria:

* Symptomatic small bowel obstruction (i.e. total parenteral nutrition, nasogastric tube).
* Previous treatment with maximum cumulative doses of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones.
* A history of allergic reaction to platinum containing compounds or doxorubicin.
* Renal impairment, defined as GFR < 40 ml/min, (Cockcroft-Gault Equation).
* Myocardial insufficiency, defined as NYHA class > 2.
* Impaired liver function defined as bilirubin ≥ 1.5 x UNL (upper normal limit).
* Inadequate hematological function defined as ANC ≤ 1.5 x 109/l and platelets ≤ 100 x109/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with major/complete histologic response (PRGS 1+2) peritoneal biopsies, within a series of three PIPAC procedures. | 4 years
  Objective Tumor response will be evaluated by the Peritoneal Regression Grading Score based on repeated peritoneal biopsies during each PIPAC procedure.

SECONDARY OUTCOMES:
Number of patients with improved Quality of Life (QoL) | 4 years
  Based on EORTC QLQC30 questionnaire at baseline and after 3 PIPAC treatments
Number of patients where MRI is accurate in describing PM distribution and progressive/regressive disease | 4 years
  Based on MRI of the abdomen at baseline and after 3 PIPAC treatments, it will be evaluated, whether MRI can detect PM and whether MRI can be used to evaluate progression/regression during PIPAC treatment. Comparative gold standard is laparoscopy including biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
Publications and presentations will be based on patient data, but the database is not open to other researchers.

REFERENCES:
- [Background] Solass W, Kerb R, Murdter T, Giger-Pabst U, Strumberg D, Tempfer C, Zieren J, Schwab M, Reymond MA. Intraperitoneal chemotherapy of peritoneal carcinomatosis using pressurized aerosol as an alternative to liquid solution: first evidence for efficacy. Ann Surg Oncol. 2014 Feb;21(2):553-9. doi: 10.1245/s10434-013-3213-1. Epub 2013 Sep 5. PMID 24006094
- [Background] Tempfer CB, Celik I, Solass W, Buerkle B, Pabst UG, Zieren J, Strumberg D, Reymond MA. Activity of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin and doxorubicin in women with recurrent, platinum-resistant ovarian cancer: preliminary clinical experience. Gynecol Oncol. 2014 Feb;132(2):307-11. doi: 10.1016/j.ygyno.2013.11.022. Epub 2013 Nov 23. PMID 24275155
- [Background] Solass W, Giger-Pabst U, Zieren J, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy (PIPAC): occupational health and safety aspects. Ann Surg Oncol. 2013 Oct;20(11):3504-11. doi: 10.1245/s10434-013-3039-x. Epub 2013 Jun 14. PMID 23765417
- [Derived] Graversen M, Lundell L, Fristrup C, Pfeiffer P, Mortensen MB. Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) as an outpatient procedure. Pleura Peritoneum. 2018 Nov 27;3(4):20180128. doi: 10.1515/pp-2018-0128. eCollection 2018 Dec 1. PMID 30911669
- [Derived] Graversen M, Detlefsen S, Asmussen J, Mahdi B, Fristrup C, Pfeiffer P, Mortensen MB. Treatment of peritoneal carcinomatosis with Pressurized IntraPeritoneal Aerosol Chemotherapy - PIPAC-OPC2. Pleura Peritoneum. 2018 Jun 9;3(2):20180108. doi: 10.1515/pp-2018-0108. eCollection 2018 Jun 1. PMID 30911656